CLINICAL TRIAL: NCT00063089
Title: Initial Safety and Pharmacokinetics Trial of Immune Globulin to Staphylococcus Aureus Capsule Polysaccharide (Altastaph) in Subjects With S. Aureus Bacteremia and Persistent Fever
Brief Title: Safety and Behavior of S. Aureus Immune Globulin Intravenous(Human), [Altastaph] in Patients With S. Aureus Bacteremia and Continuing Fever
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nabi-1407
Record Dates: First submitted 2003-06-19; First posted 2003-06-20 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Staphylococcal Infections
Keywords: Staphylococcal infection; Gram positive bacteria; Staphylococcus; Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- altastaph (Experimental): S. aureus Immune Globulin Intravenous (Human) 5%
  Interventions: Drug: S. aureus Immune Globulin Intravenous (Human) 5%
- Placebo (Placebo Comparator): 0.45% Normal Saline
  Interventions: Drug: S. aureus Immune Globulin Intravenous (Human) 5%

INTERVENTIONS:
Drug: S. aureus Immune Globulin Intravenous (Human) 5%

SUMMARY:
Altastaph has been developed to help the removal of S. aureus from the bloodstream. The main objective of this study will be to test the safety and behavior of Altastaph in patients with S.aureus bacteremia and continuing fever

DETAILED DESCRIPTION:
Staphylococcus aureus has been recognized as an important community - acquired and nosocomial pathogen. Because it is a common cause of osteomyelitis, endocarditis, and meningitis, S. aureus infections lead to considerable morbidity and mortality. The main objective of this study will be to test the safety and pharmacokinetics of Altastaph in patients with S. aureus bacteremia and persistent fever. This study will also assess the efficacy of Altastaph versus control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 7 years of age
* Weight less then or equal to 150 kilograms
* Subjects willing to complete the full duration of the study, including the follow up visit to day 42
* Life expectancy will enable the subject to complete the duration of the study
* Female subjects of child-bearing potential, negative serum pregnancy test prior to the first infusion of study material. Female subjects of child-bearing potential must agree to use an effective method of birth control throughout the study. Abstinence is not considered an adequate birth control measure. Female subjects of non-child-bearing potential must have history of hysterectomy, bilateral surgical or radiation-induced oophorectomy, tubal ligation or evidence of post menopausal status
* Subject, legal guardian(s) or medical power of attorney must have given written informed consent/ assent
* S. aureus bacteremia and persistent fever. S. aureus bacteremia is defined as the first blood culture positive for S. aureus (index blood culture). Persistent fever (qualifying fever) is defined as a temperature (greater then or equal to 100.4F or greater then or equal to 38C) occuring at least 24 hours after the index temperature was recorded and after the index blood culture was drawn
* Absolute Neutrophil Count (ANC) greater then or equal to 500 x 10^9 cells/L
* Subjects with malignancies may participate if:(1) The malignancy is a solid tumor (i.e. not lymphoma, leukemia, etc.)(2) The tumor has not metastasized to the bone marrow

Exclusion Criteria:

* Known hypersensitivity or previous anaphylaxis to polysaccharide or polysaccharide-conjugate vaccines or to any component of Altastaph
* Profound disability, assessed by the investigator, which would prevent participation in the study
* Known IgA deficiency
* Known HIV infection with CD4 count < 200 cells/L
* Presence of any conditions which, in the opinion of the investigator, places the subject at undo risk or potentially jeopardizes the quality of the data to be generated
* Pregnancy or breast feeding
* Use of investigational drug or biologic in the four weeks prior to screening and during the study. The only exception is use of investigational antineoplastic product if, and only if: (1) The product is not expected to result in sever and prolonged immunosuppression (2) The product is, itself, not immunologically-based (e.g. anti-tumor/ monoclonal antibodies, cancer vaccines or interleukins

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-09; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Safety | 6 weeks

SECONDARY OUTCOMES:
pharmacokinetics | 6 weeks
Efficacy | 6 Weeks

REFERENCES:
- [Derived] Rupp ME, Holley HP Jr, Lutz J, Dicpinigaitis PV, Woods CW, Levine DP, Veney N, Fowler VG Jr. Phase II, randomized, multicenter, double-blind, placebo-controlled trial of a polyclonal anti-Staphylococcus aureus capsular polysaccharide immune globulin in treatment of Staphylococcus aureus bacteremia. Antimicrob Agents Chemother. 2007 Dec;51(12):4249-54. doi: 10.1128/AAC.00570-07. Epub 2007 Sep 24. PMID 17893153